CLINICAL TRIAL: NCT05189951
Title: The Effect of Different Wiping Motions in Phlebotomy on Vein Visibility, Procedural Success and Phlebotomy-related Complications
Brief Title: Different Wiping Motions in Phlebotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Instructor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 817
Record Dates: First submitted 2021-12-21; First posted 2022-01-13 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Nurse's Role

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- circular motion (Experimental): The phlebotomy site was wiped in a circular motion from the center outwards, approximately 5x5 cm wide.
  Interventions: Other: circular motion
- vertical motion (Experimental): The phlebotomy site was wiped vertically from top to bottom with a single maneuver.
  Interventions: Other: vertical motion
- first vertical then circular motion (Experimental): The phlebotomy site was first vertically wiped from top to bottom with a single maneuver, and then it was wiped in a circular motion from the center to the outside. Different swabs were used in both wipes.
  Interventions: Other: circular+vertical motion

INTERVENTIONS:
Other: circular motion — The phlebotomy site was wiped in a circular motion from the center outwards, approximately 5x5 cm wide.
  Arms: circular motion
Other: vertical motion — The phlebotomy site was wiped vertically from top to bottom with a single maneuver.
  Arms: vertical motion
Other: circular+vertical motion — The phlebotomy site was first vertically wiped from top to bottom with a single maneuver, and then it was wiped in a circular motion from the center to the outside.
  Arms: first vertical then circular motion

SUMMARY:
This study was conducted with 90 patients. The phlebotomy site was wiped with circular motion in the group-I, vertical movement in the group-II, and first vertical and then circular motion in the group-III.

DETAILED DESCRIPTION:
Aim: This study was conducted to evaluate the effects of different wiping motions used in phlebotomy on vein visibility, procedural success, and phlebotomy-related complications.

Background: In phlebotomy practice, many application guidelines or textbooks are used. In these references, it is seen that phlebotomy site is wiped with different motions.

Methods: This study was conducted with 90 patients. The phlebotomy site was wiped with circular motion in the group-I, vertical movement in the group-II, and first vertical and then circular motion in the group-III.

ELIGIBILITY:
Inclusion Criteria:

* who are over 18 years old,
* without any psychiatric diseases,
* without vision or hearing problems,
* hospitalized in the internal medicine clinic,
* with platelet counts of 200 000 / mm³ and above,
* 8 cc of blood is ordered for lab test and
* individuals who volunteered to participate in the study

Exclusion Criteria:

* having a local or systemic infection,
* having vascular disease,
* having an immunopathological problem,
* scarring, psoriasis, active dermatitis in the phlebotomy site,
* having peripheral nerve disease,
* having peripheral neuropathy,
* patients with coagulation disorder,
* individuals who don't volunteered to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Vein Assessment | up to 1 minute after wiping the venipuncture site
  This evaluation has a total of 5 assessment steps, (1) veins are neither visible nor palpable, (2) veins are visible but not palpable, (3) veins are barely visible and palpable, (4) veins are visible and palpable, and (5) veins are clearly visible and easily palpable.
Change in complications at 72 hours | 24th, 48th and 72nd hour
  The results of evaluations such as complication development and size of the complications. It was evaluated three times at the 24th, 48th and 72nd hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)